CLINICAL TRIAL: NCT02219906
Title: Resveratrol in Metabolic Syndrome: Effect on Platelet Hyper-reactivity and HDL Lipid Peroxidation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, John Oates, Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 130996
Record Dates: First submitted 2014-08-14; First posted 2014-08-19 (Estimated); Last update posted 2019-04-19 (Actual); Status verified 2019-04

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome | interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo capsule given three times daily X 3 weeks
  Interventions: Dietary Supplement: Placebo
- Resveratrol (Experimental): Resveratrol 1 gram three times daily X 3 weeks
  Interventions: Dietary Supplement: Resveratrol

INTERVENTIONS:
Dietary Supplement: Resveratrol — 1000mg tid
  Other Names: tid dosing
  Arms: Resveratrol
Dietary Supplement: Placebo — 1000mg tid placebo
  Other Names: tid dosing
  Arms: Placebo

SUMMARY:
Metabolic syndrome is a group of risk factors that increase a patient's likelihood for heart attack, stroke and diabetes. Our research is aimed at understanding whether a drug, resveratrol, commonly found in grapes and red wine, would have any benefit in reducing risk factors in patients that have metabolic syndrome. Despite the use of aspirin and cholesterol reducing medications, patients with metabolic syndrome still often have sticky platelets and dysfunctional lipid profile. This is likely due to inflammation and high oxidative state. In animal studies, this drug has reduced platelet stickiness and reduced oxidative stress. However, the effects of this drug have not been researched in patients with metabolic syndrome.

We are interested in studying whether the benefits of resveratrol described in animal models can be translated to patients with metabolic syndrome who display high markers of oxidative stress. We plan to give a short intervention of drug to patients and then determine if the drug successfully:

1. Decreases the stickiness of platelets. This is important because sticky platelets are more likely to form clot and contribute to plaque formation.
2. Reduce the circulating dysfunctional HDL. HDL and its protein and lipid constituents help to inhibit oxidation, inflammation, activation of the blood vessel wall, coagulation, and platelet aggregation. Dysfunctional HDL, as occurs in metabolic syndrome patients, cannot properly protect against atherosclerosis.

DETAILED DESCRIPTION:
Patients with metabolic syndrome are at increased risk of thrombotic complications, including myocardial infarction and cardiovascular death. A meta-analysis of the studies assessing cardiovascular risk in metabolic syndrome found a pooled relative risk for incident cardiovascular events and death of 1.78. This propensity for thrombotic vascular events is in the context of an increasing prevalence of metabolic syndrome, which in the 2003-2006 NHANES Survey was found in 34% of the US population over the age of 20.

Two important contributors to the development of myocardial infarction and stroke are lipid rich atheromatous plaques and concomitant platelet aggregation in response to the fissuring of these plaques. A growing body of evidence implicates oxidative modification of lipoprotein lipids and apolipoproteins in the genesis of plaques. Platelet hyperactivity and the variable response to antiplatelet therapy are features of the metabolic syndrome. Oxidative modifications of LDL enhance activation of platelets, which themselves are oxidatively stressed. Myeloperoxidase (MPO) initiates lipid peroxidation leading to dysfunctional HDL production. Therefore, the hypotheses for the proposed investigations will address the effects of resveratrol on platelet hyperactivity and HDL protein modifications in patients with metabolic syndrome. Resveratrol, as predicted from its structure, is an electron rich molecule that can reduce free radicals. It has distinctive actions, however, that differ from compounds that are conventionally referred to as "anti-oxidants". It has particular potency as an inhibitor of radical formation by a number of peroxidases that likely participate in the pathophysiology of metabolic syndrome. These include MPO, the peroxidase site of prostaglandin H synthase-1 (PGHS-1; cyclooxygenase-1(COX-1)) and cytochrome c.

We will test the hypothesis that:

1. resveratrol reduces platelet activation in patients with metabolic syndrome. and
2. that resveratrol reduces the oxidative modification of HDL proteins in patients with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Metabolic Syndrome

Exclusion Criteria:

* Evidence of coronary artery disease
* Indication for use of aspirin for secondary prevention of thrombotic events
* Use of non-steroidal anti-inflammatory drugs or anti-platelet agents
* Pregnancy
* Patients with history of bleeding or gastrointestinal ulcers
* Patients with major illnesses such as ongoing malignancies, infections, cirrhosis

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-05; Primary Completion 2019-02-07 (Actual); Study Completion 2019-04-07 (Actual)

PRIMARY OUTCOMES:
Change in parameters of platelet activation | baseline, 3 weeks after intervention
  Measure platelet-monocyte aggregates by flow cytometry
Change in parameter for platelet oxidative stress | Baseline, 3 weeks after intervention
  Measure malondialdehyde adducts of platelet proteins
Change in parameter for platelet oxidation levels | Baseline, 3 week after intervention
  Measure superoxide production by platelets
Serum Thromboxane measurments | Baseline, 3 weeks after intervention
  Measure thromboxane to assess inflammation

SECONDARY OUTCOMES:
Change in oxidative modifications of HDL | baseline, three weeks after intervention
  Measure change in malondialdehyde adducts in HDL proteins
Change in plasma oxidative stress | baselines, three weeks after intervention
  Measure change in plasma isoprostanes

CONTACTS AND LOCATIONS:
Overall Officials: John A Oates, MD, Principal Investigator — Vanderbilt University
Locations (2):
- United States (2):
  - Vanderbilt University, Nashville, Tennessee
  - Baylor University, Houston, Texas

IPD SHARING:
Plan to Share IPD: No